CLINICAL TRIAL: NCT05043883
Title: Automated Assessment of Pulmonary Vein Isolation (PVI) Using a Novel EP Recording System (CathVision Cube® System)
Brief Title: Automated Assessment of PVI Using a Novel EP Recording System
Acronym: PVISION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CathVision ApS (Industry)
Collaborators: AKRN Scientific Consulting, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPVI-002
Record Dates: First submitted 2021-08-03; First posted 2021-09-14 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: atrial fibrillation; pulmonary vein isolation; radiofrequency; cryo balloon; ablation; software; pulse field ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental): Index EP Procedure: Ablation of atrial fibrillation
  Interventions: Device: CathVision Cube® system

INTERVENTIONS:
Device: CathVision Cube® system — Intracardiac signals will be passively recorded using the investigational CathVision Cube® System in parallel with the commercial (bearing CE mark) EP recording systems LabSystem Pro, Boston Scientific EP, or EP-Tracer, Schwarzer Cardiotek. The investigational device will not be used for direct clinical care decisions or therapy. The validation of the PVI Analyzer will be performed offline and retrospectively.

SUMMARY:
A prospective, multi-center study with the CathVision Cube® system and the PVI Analyzer software in radiofrequency (RF), cryo-balloon (CB), and Pulse Field Ablation (PFA) procedures.

DETAILED DESCRIPTION:
Subjects with paroxysmal or persistent atrial fibrillation (AF) who are indicated to undergo first pulmonary vein isolation (PVI) procedure and meet all eligibility criteria will be enrolled in the Study. Intracardiac signals will be passively recorded using the investigational CathVision Cube® System in parallel with the conventional (CE marked) EP recording system. The investigational device will not be used for direct clinical care decisions or therapy. The validation of the automated algorithm for PVI will be performed offline

The primary objective is to validate the PVI Analyzer software with a novel EP recording system (CathVision Cube® System) for assisting assessment of isolation status following PVI ablation.

The secondary objective is to determine the feasibility of "real-time" assessment of PVI analysis and rhythm dependent performance using the PVI Analyzer and CathVision Cube® System.

ELIGIBILITY:
Eligible subjects will meet all of the following inclusion criteria:

1. Subjects undergoing first-time pulmonary vein isolation indicated by investigator for the treatment of atrial fibrillation
2. Male or non-pregnant female aged ≥21 years.
3. Able and willing to provide written informed consent prior to any clinical investigation related procedure

Eligible subjects will not meet any of the following exclusion criteria:

1. Pregnant or nursing subjects.
2. Current participation in another investigational drug or device study that interferes with this Study.
3. Subjects who, in the opinion of the investigator, are not candidates for this Study.
4. Patients who have had a prior ablation procedure
5. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
6. Life expectancy less than 12 month
7. Subjects who, in the opinion of the investigator, are considered part of any vulnerable population.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Duytschaever, Prof. MD PhD, Principal Investigator — AZ Sint-Jan Hospital, Ruddershove 10 8000 Brugge, Belgium
Locations (4):
- Belgium (3):
  - AZ Sint-Jan Hospital, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Ghent University Hospital, Ghent
- Clinique Pasteur Toulouse,, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment took place between September 15, 2021 and June 22, 2022 at four sites (hospitals) located in Bruges, Brussels, Ghent and Toulouse. At these hospitals, participants were assessed for eligibility to participate in the clinical investigation, and those who met the eligibility criteria, voluntarily gave their informed consent. Those who were successfully enrolled were monitored until their hospital discharge, and no further follow-up was deemed necessary.
Pre-assignment Details: Three of the subjects were considered screening failures since not all eligibility criteria were met, and the subjects were excluded from the study. Out of the 101 subjects enrolled, 4 subjects were excluded from the Per-Protocol Treatment analysis, as minimum required measurements could not be taken. Therefore, the final PPT population for analysis was 97 subjects.
Groups:
- Index EP Procedure: Ablation of Atrial Fibrillation: This is a single arm study that is assigned to subjects undergoing first-time pulmonary vein isolation indicated by investigator for the treatment of atrial fibrillation. Subjects were distributed in two different procedures (RF and cryo-balloon) according to medical decision and standard of care practice at the study sites. At a later stage, a protocol amendment planned an additional enrolment undergoing the standard of care PFA procedure
  Intracardiac signals will be passively recorded using the investigational CathVision Cube® System in parallel with the commercial (bearing CE mark) EP recording systems LabSystem Pro, Boston Scientific EP, or EP-Tracer, Schwarzer Cardiotek. The investigational device will not be used for direct clinical care decisions or therapy. The validation of the PVI Analyzer will be performed offline and retrospectively.
Period: Overall Study
Arm/Group | Index EP Procedure: Ablation of Atrial Fibrillation
Started | 101 (The total number of consented patients was 104; however, three of them did not meet the eligibility criteria and were classified as screening failures. Therefore, 101 subjects were successfully enrolled in this clinical investigation.)
Completed | 97 (Subjects may be classified in either the Intent-to-Treat (ITT) or Per-Protocol Treatment (PPT) populations, as defined in the clinical investigation plan. Out of the 101 subjects enrolled in this clinical investigation, 4 subjects were excluded from the PPT analysis. Minimum required measurements as per the Statistical Analysis Plan (SAP) could not be taken)
Not Completed | 4
Not completed — Minimum required measurements could not be taken | 4

BASELINE CHARACTERISTICS:
Groups:
- Index EP Procedure: Ablation of Atrial Fibrillation: CathVision Cube® system: Intracardiac signals will be passively recorded using the investigational CathVision Cube® System in parallel with the commercial (bearing CE mark) EP recording systems LabSystem Pro, Boston Scientific EP, or EP-Tracer, Schwarzer Cardiotek. The investigational device will not be used for direct clinical care decisions or therapy. The validation of the PVI Analyzer will be performed offline and retrospectively.
Arm/Group | Index EP Procedure: Ablation of Atrial Fibrillation
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.76 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [cm] [Mean (Standard Deviation); unit: cm] | 174.23 (9.83)
Weight [kg] [Mean (Standard Deviation); unit: kg] | 82.04 (17.86)
Systolic Blood Pressure [mmHg] [Mean (Standard Deviation); unit: mmHg] | 137.39 (20.04)
Diastolic Blood Pressure [mmHg] [Mean (Standard Deviation); unit: mmHg] | 79.44 (12.10)
Heart Rate [BPM] [Mean (Standard Deviation); unit: BPM] | 72.69 (22.40)
Respiratory Rate [breaths/min] [Mean (Standard Deviation); unit: breaths/min] | 14.88 (5.17)
Body Temperature [°C] [Mean (Standard Deviation); unit: ºC] | 36.28 (0.42)

OUTCOME MEASURES:

1. Primary Outcome: PVI Analyzer Sensitivity and Specificity, Measured as the Accuracy of Predictions for Non-isolated and Isolated Veins.
Description: The primary outcome is to evaluate the sensitivity and specificity of the PVI Analyzer in the classification of the isolation status of veins, following the medical procedure known as pulmonary vein isolation (PVI). The information used for this has been obtained from the investigational CathVision Cube System. The PVI Analyzer determines whether the veins are isolated or not after pulmonary vein ablation.
  The proportion of correct negative (non-isolated) predictions among non-isolated vein data points and the proportion of correct positive (isolated) data points from isolated veins, provide the sensitivity and specificity data, respectively.
Time Frame: From EP procedure until study completion at discharge; an average of 24 hours.
Population: The performance assessment was done in the PPT population, with a total of 85 subjects. Subjects undergoing PFA were excluded from this analysis despite being included in the PPT population, since the primary endpoint was specific to RF and Cryo procedures only.
  Up to 248 EGMs were recorded at 'T-baseline' (prior to isolation) and labeled as ground-truth negative (non-isolated); and 250 EGMs were recorded at 'T-final' (after isolation) and labeled as ground-truth positive (isolated).
Measure: Count of Units; unit: Electrogram (EGM)
Units Other Than Participants: Electrogram (EGM)
Arm/Group | Single Group
Number analyzed (Participants) | 85
Number analyzed (Electrogram (EGM)) | 498
Electrogram (EGM)
  Sensitivity: number analyzed (Electrogram (EGM)) | 250
  Sensitivity | 216
  Specificity: number analyzed (Electrogram (EGM)) | 248
  Specificity | 215
Statistical Analysis 1: Comparison: Single Group; Specificity is the ability to correctly detect true negative values of the ground-truth negative EGM classifications. The PVI Analyzer software classifies an EGM in positive (isolated) or negative (non-isolated), compared to the SOC outcomes. EGMs prior-isolation were labeled as ground-truth negative (non-isolated), EGMs after isolation as ground-truth positive (isolated). The null hypothesis is that specificity is lower or equal to the superiority limit 80%; Test type: Superiority — This clinical investigation is intended to demonstrate that the performance of the PVI Analyzer software is superior to clinically relevant performance level, and therefore the study is designed as a 1-sample superiority test of the sampled outcome specificity. The lower bound 95% CI (α=0.05) and at a statistical power of 95% (β=0.05); p = 0.006, Z-test — The success of the PVI Analyzer output was assumed to follow a binominal distribution with a given true proportion of 87.50%. It was tested whether the specificity was superior to the 80% limit; A one-tailed test with a significance level of 95% (α = 0.05) was applied; Percentage (%) = 87
Statistical Analysis 2: Comparison: Single Group; Sensitivity of the PVI analyzer is determined by the capability to detect true positive among all ground-truth positive EGM classifications.The PVI Analyzer software classifies an EGM in positive (isolated) or negative (non-isolated), compared to the SOC outcomes. EGMs prior-isolation were labeled as ground-truth negative (non-isolated), EGMs after isolation as ground-truth positive (isolated). The null hypothesis is that sensitivity is lower or equal to the superiority limit 80%; Test type: Superiority — This clinical investigation is intended to demonstrate that the performance of the PVI Analyzer software is superior to clinically relevant performance level, and therefore the study is designed as a 1-sample superiority test of the sampled outcome Sensitivity. The lower bound 95% CI (α=0.05) and at a statistical power of 95% (β=0.05); p = 0.004, Z-test — The success of the PVI Analyzer output was assumed to follow a binominal distribution with a given true proportion of 87.50%. It was tested whether the sensitivity was superior to the 80% limit; A one-tailed test with a significance level of 95% (α = 0.05) was applied; Percentage = 86

2. Primary Outcome: PVI Analyzer Safety Profile, Measured as the Number of Adverse Events and/or Device Malfunctions.
Description: As part of the primary outcome, safety is also evaluated as the number of adverse events and device malfunctions reported by the study team at site, during the use of the CathVision Cube® System from the start of the procedure until discharge. The number of adverse events and device malfunctions is recorded in the site's source documents as well as in the case report form (CRF) and is duly informed to the Sponsor who also keeps the record.
Time Frame: From EP procedure until study completion at discharge; an average of 24 hours.
Population: All enrolled subjects.
Measure: Number; unit: participants
Arm/Group | Single Group
Number analyzed (Participants) | 101
participants
  Mild | 0
  Moderate | 1
  Severe | 0
  Device related | 0
  Procedure related | 1
  other | 0
  Serious Adverse Events | 1
  Serious adverse device effect (SADE) incidence | 0
  Serious unanticipated serious adverse device effect (USADE) incidence | 0
  Device deficiency incidence | 0
Statistical Analysis 1: Comparison: Single Group; A descriptive analysis was performed to evaluate the AEs and device deficiencies, estimating the percentages and 95% CI on each category; Test type: Other — Descriptive; Percentage = 0.99, 95% CI 2-sided [0.02 to 5.39], Standard Deviation 0.10 — Only one AE was reported for one subject ( which was considered moderate in severity and not related to the device, but related to the SOC procedure

3. Secondary Outcome: The Pulmonar Vein Isolation (PVI) Classification in Sinus Rhythm (SR) Considering the Electrophysiology Procedure Type.
Description: This outcome assesses the overall classification of pulmonary vein isolation (PVI) in sinus rhythm (SR) based on the type of electrophysiology procedure performed. The classification provides insights into the accuracy of the procedure in achieving SR.
  The overall classification was evaluated in terms of sensitivity and specificity. To calculate specificity from the total number of EGMS analyzed, all the correct negatives (non-isolated) / Correct negatives + False positives were considered. To calculate sensitivity, all the correct positives (isolated) / Correct positives + False negatives were considered.
  As the sample size was not adjusted to detect the differences for variables other than the primary endpoint, the p-values obtained from the analyses of secondary outcomes should be viewed as complementary to the primary outcome results. Their primary purpose was to generate hypotheses rather than draw definitive conclusions.
Time Frame: From EP procedure until study completion at discharge; an average of 24 hours.
Population: This secondary outcome assessed the overall classification accuracy of the PVI Analyzer in sinus rhythm (SR) computing the results only in radiofrequency and cryoballoon procedures. Therefore, the dataset used for the analysis is the same as for the primary endpoint (85), but subgrouping the data by the type of procedure.
Measure: Count of Units; unit: Electrogram (EGM)
Units Other Than Participants: Electrogram (EGM)
Groups:
- Radiofrequency Procedure: Index EP Procedure: Ablation of atrial fibrillation according to Radiofrequency Procedure: Radiofrequency delivery ablates the tissue through heat.
  CathVision Cube® system: Intracardiac signals will be passively recorded using the investigational CathVision Cube® System in parallel with the commercial (bearing CE mark) EP recording systems LabSystem Pro, Boston Scientific EP, or EP-Tracer, Schwarzer Cardiotek. The investigational device will not be used for direct clinical care decisions or therapy. The validation of the PVI Analyzer will be performed offline and retrospectively.
- Cryoballoon Procedure: Index EP Procedure: Ablation of atrial fibrillation according to Cryo-ballon Procedure: cryo-balloon ablates the tissue through freezing.
  CathVision Cube® system: Intracardiac signals will be passively recorded using the investigational CathVision Cube® System in parallel with the commercial (bearing CE mark) EP recording systems LabSystem Pro, Boston Scientific EP, or EP-Tracer, Schwarzer Cardiotek. The investigational device will not be used for direct clinical care decisions or therapy. The validation of the PVI Analyzer will be performed offline and retrospectively.
- Pulsed Field Ablation (PFA) Procedure: PFA delivers short high-voltage pulses that ablates through irreversible electroporation.
  The data obtained from pulsed field ablation (PFA) analysis could not be assessed for this secondary endpoint as it was found to be incompatible with the PVI Analyzer algorithm, which requires the PV mapping catheter to have eight or ten electrodes and the PFA catheter has only five.
Arm/Group | Radiofrequency Procedure | Cryoballoon Procedure | Pulsed Field Ablation (PFA) Procedure
Number analyzed (Participants) | 42 | 47 | 12
Number analyzed (Electrogram (EGM)) | 258 | 240 | 0
Electrogram (EGM)
  Specificty: number analyzed (Electrogram (EGM)) | 127 | 121 | 0
  Specificty | 120 | 95 | 0
  Sensitivity: number analyzed (Electrogram (EGM)) | 131 | 119 | 0
  Sensitivity | 107 | 109 | 0
Statistical Analysis 1: Comparison: Radiofrequency Procedure; Automated PVI Analyzer classification of PV isolation in SR by Radiofrequency procedure from EP procedure until study completion at discharge (an average of 24 hours), with a specificity superior to 80%. A superiority Z-test for Specificity was performed; Test type: Superiority; p = 0.00002, Z-test — Computed p values are the result of running a one sample z-test with a null hypothesis that specificity is below 80%; Percentage (%) = 94
Statistical Analysis 2: Comparison: Radiofrequency Procedure; Automated PVI Analyzer classification of PV isolation in SR by Radiofrequency procedure from EP procedure until study completion at discharge (an average of 24 hours), with sensitivity superior to 80%. A superiority Z-test for Sensitivity was performed; Test type: Superiority; p = 0.32, Z-test — Computed p values are the result of running a one sample z-test with a null hypothesis that sensitivity is below 80% and alternative hypothesis that sensitivity is at or above 80%; Percentage (%) = 82
Statistical Analysis 3: Comparison: Cryoballoon Procedure; Automated PVI Analyzer classification of PV isolation in SR by Cryo-balloon procedure from EP procedure until study completion at discharge (an average of 24 hours), with a specificity superior to 80%. A superiority Z-test for Specificity was performed; Test type: Superiority; p = 0.66, Z-test — Computed p values are the result of running a one sample z-test with a null hypothesis that specificity is below 80%; Percentage (%) = 79
Statistical Analysis 4: Comparison: Cryoballoon Procedure; Automated PVI Analyzer classification of PV isolation in SR by Cryo-balloon procedure from EP procedure until study completion at discharge (an average of 24 hours), with a sensitivity superior to 80%. A superiority Z-test for Sensitivity was performed; Test type: Superiority; p = 0.0008, Z-test — [p-value comment as in outcome 3, analysis 2]; Percentage (%) = 92

4. Secondary Outcome: Feasibility of "Real-time" Assessment of Isolation, Measured by Retesting the Accuracy of the PVI Analyzer Classification of Isolation Status at Different Timepoints Before, During and After Ablation.
Description: The device's feasibility was evaluated by reassessing its accuracy. It refers to the consistency in the re-classification of pairs of non-overlapping samples throughout the different timepoints of ablation-prior to, during, and following the procedure. For this evaluation, the same EGMs of the primary endpoint were used, including only EGMs from T Baseline and T Final measurements from patients in sinus rhythm.
  The extraction of non-overlapping samples was selected by considering only those EGMs with a number of global isolation index values above 6. The global isolation index value is an indicator from the PVI analyzer that is used to assess the overall effectiveness of the ablation in isolating specific regions of the heart. The fourth and last global index returned by the PVI Analyzer were used as pairs for analyzing the outcome.
  The accuracy was calculated as the percentage of EGMs with agreement across timepoints with respect to the total number of EGMs performed.
Time Frame: From EP procedure until study completion at discharge; an average of 24 hours.
Population: EGMs with a number of global isolation index values above 6 were selected. For those EGMs, the fourth and last global index returned by the PVI Analyzer were used. This value was compared at different time points of the procedure, to confirm whether there was an ECG agreement or not. The number of EGM with agreement was 475/495, and the number of EGM without agreement was 20/475.
Measure: Count of Units; unit: Electrogram (EGM)
Units Other Than Participants: Electrogram (EGM)
Arm/Group | Index EP Procedure: Ablation of Atrial Fibrillation
Number analyzed (Participants) | 85
Number analyzed (Electrogram (EGM)) | 495
Electrogram (EGM) | 475
Statistical Analysis 1: Comparison: Index EP Procedure: Ablation of Atrial Fibrillation; This endpoint used the same EGMs extracted for the primary endpoint, including only EGMs from T Baseline and T Final measurements from patients in sinus rhythm; Test type: Superiority; p = 0.000005, Z-test — To compute the proportional agreement between two non-overlapping samples, a one-sample Z-test was performed with the alternative hypothesis that agreement was above 90%, which was considered sufficient for a real-time assessment; Percentage (%) = 96

5. Secondary Outcome: PVI Isolation Classification in Non-sinus Rhythm (NSR) From EP Procedure
Description: The PVI isolation classification in non-sinus rhythm (NSR) from EP procedure was focused on the analysis of all EGM in non-sinus rhythm. The data analysis and processing were similar to those of the primary endpoint, but taking into consideration that subjects shall be in non-sinus rhythm during the duration of the EGM snippet.
  Apart from this, the processing was the same and the threshold was also defined as 50: values below 50 were classified as baseline, while values at or above 50 were considered as isolated veins.
Time Frame: From EP procedure until study completion at discharge; an average of 24 hours.
Population: The performance assessment was done in the Per Protocol (PPT) population, with a total of 85 participants. The PVI isolation classification in non-sinus rhythm (NSR) from EP procedure was focused on the analysis of all EGM in non-sinus rhythm which in this case were 55 in T-baseline and 44 in T-final, a total of 99 ECGs. However, the system rejected 9 ECGs in T-baseline and 3 in T-final, therefore, the ECGs used for this secondary outcome were 46 in T-baseline and 41 in T-final.
Measure: Count of Units; unit: Electrogram (EGM)
Units Other Than Participants: Electrogram (EGM)
Arm/Group | Index EP Procedure: Ablation of Atrial Fibrillation
Number analyzed (Participants) | 85
Number analyzed (Electrogram (EGM)) | 87
Electrogram (EGM)
  Specificity: number analyzed (Electrogram (EGM)) | 46
  Specificity | 25
  Sensitivity: number analyzed (Electrogram (EGM)) | 41
  Sensitivity | 41
Statistical Analysis 1: Comparison: Index EP Procedure: Ablation of Atrial Fibrillation; The data analysis and processing were similar to those of the primary endpoint, but taking into consideration that subjects shall be in non-sinus rhythm during the duration of the EGM snippet. Apart from this, the processing was the same and the threshold was also defined as 50: values below 50 were classified as baseline, while values at or above 50 were considered as isolated veins; Test type: Superiority; p = 1, Z-test — The p values calculated are the result of running a one sample z-test with a null hypothesis that the specificity are below 80%; Percentage (%) = 54
Statistical Analysis 2: Comparison: Index EP Procedure: Ablation of Atrial Fibrillation; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0007, Z-test — The p values calculated are the result of running a one sample z-test with a null hypothesis that the sensitivity are below 80% and an alternative hypothesis that sensitivity is at or above 80%; Percentage (%) = 100

6. Secondary Outcome: Accuracy of PVI Analyzer Classification at the Time of Expert-defined Isolation
Description: This secondary endpoint aimed to determine the sensitivity of the PVI Analyzer at the time of isolation, which requires the EGMs at the T PVI. The T PVI EGMs were extracted by taking EGM snippets of 4 seconds around the T PVI event. All of those EGMs were expected to be from isolated veins (ground-truth is isolated). Then, they were processed by the PVI Analyzer, and the last valid global isolation index output was used for endpoint assessment.
Time Frame: From EP procedure until study completion at discharge; an average of 24 hours.
Population: In many cases, the actual isolation time was not directly observable, and the investigator was only asked to annotate T PVI if it was observed.
  During RF procedures, T PVI can be difficult to observe and during cryo-balloon application, freeze noise from the cryoballoon can make identification of T PVI difficult. The annotation the EGMs at the T PVI was not always possible and only 116 valid EGMs at T PVI were collected. During processing, 17 EGMs were rejected by the PVI Analyzer.
Measure: Count of Units; unit: Electrogram (EGM)
Units Other Than Participants: Electrogram (EGM)
Arm/Group | Index EP Procedure: Ablation of Atrial Fibrillation
Number analyzed (Participants) | 85
Number analyzed (Electrogram (EGM)) | 99
Electrogram (EGM) | 86
Statistical Analysis 1: Comparison: Index EP Procedure: Ablation of Atrial Fibrillation; This secondary endpoint aimed to determine the sensitivity of the PVI Analyzer at the time of isolation, which requires the EGMs at the T PVI. A Z-test for sensitivity was performed to assess the sensitivity of the PVI Analyzer analysis to identify expert-defined isolation during the PVI ablation; Test type: Superiority; p = 0.04, Z-test; The estimate was done using a one-sample Z-test with a null hypothesis that sensitivity is at or below 80% and a 95% significance level; Percentage (%) = 87

7. Secondary Outcome: Comparison of the PVI Analyzer Performance With CathVision Cube® System Data With Its Performance With Data From Other Conventional EP Systems Used
Description: The conventional EP system and CathVision Cube® System were running on two different PCs in the EP laboratory in parallel. The relevant EGM snippets were extracted from the conventional EP system using a time offset between the conventional EP system PC and the Cube PC. Since a very similar number of samples were used to compute the results, no statistical assessment of the sampling variation in the sensitivity and specificity was made. A paired McNemars test, with an alpha value of 0.05, was applied to analyze the differences in classification performance.
Time Frame: From EP procedure until study completion at discharge; an average of 24 hours.
Population: It was not possible to extract all EGM snippets from the conventional systems, as all data from Toulouse was not available. Due to technical reasons and time constraints, only the first 12 patients from Ghent were included in the analysis.
Measure: Count of Units; unit: Electrogram (EGM)
Units Other Than Participants: Electrogram (EGM)
Groups:
- Conventional EP System: EP-Tracer, Schwarzer Cardiotek EP tracer anonymized binary files containing EGM data and event annotations, can be directly accessed in Python and processed by the PVI Analyzer.
  Boston Scientific LSPro LS Pro data is exported manually as anonymized ASCII files using the LS Pro software. All relevant pages are exported. The ASCII files can be read in Python and processed by the PVI Analyzer
- CathVision Cube® System: PVI Analyzer software used with the novel EP recording system
Arm/Group | Conventional EP System | CathVision Cube® System
Number analyzed (Participants) | 12 | 12
Number analyzed (Electrogram (EGM)) | 297 | 295
Electrogram (EGM)
  Specificity: number analyzed (Electrogram (EGM)) | 148 | 148
  Specificity | 118 | 127
  Sensitivity: number analyzed (Electrogram (EGM)) | 149 | 147
  Sensitivity | 103 | 124
Statistical Analysis 1: Comparison: Conventional EP System vs CathVision Cube® System; A paired McNemar's Chi-Square test was performed to analyze the differences in classification performances; Test type: Other; p = 0.0002, McNemars test — McNemar test assumes as a null hypothesis that the two datasets cause the PVI Analyzer to have a similar proportion of errors; A paired McNemars test with an alpha value of 0.05, was applied to analyze the differences in classification performance

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from participants' electrophysiology procedure until study completion at discharge (hospitalization time approximately 1-2 days).
Description: The assessment of the PVI Analyzer software analysis was performed offline and retrospectively, the AEs related to the device and device malfunctions reported were expected to be minimal or even absent. Determination of whether the investigational product contributed to an AE is to be determined by the Investigator. All efforts were made by the investigator to remain alert to possible AEs.
Groups:
- Adult Patients With Cardiac Arrhythmia Undergoing Cryoballoon: Safety was evaluated in adult patients diagnosed with cardiac arrhythmia, including patients with supraventricular tachycardia and ventricular tachycardia undergoing Cryoballoon procedure
- Adult Patients With Cardiac Arrhythmia Undergoing Radiofrequency: Safety was evaluated in adult patients diagnosed with cardiac arrhythmia, including patients with supraventricular tachycardia and ventricular tachycardia undergoing Radiofrequency procedure
- Adult Patients With Cardiac Arrhythmia Undergoing Pulsed Field Ablation: Safety was evaluated in adult patients diagnosed with cardiac arrhythmia, including patients with supraventricular tachycardia and ventricular tachycardia undergoing Pulsed Field Ablation procedure
Arm/Group | Adult Patients With Cardiac Arrhythmia Undergoing Cryoballoon | Adult Patients With Cardiac Arrhythmia Undergoing Radiofrequency | Adult Patients With Cardiac Arrhythmia Undergoing Pulsed Field Ablation
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/42 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/47 | 1/42 | 0/12
Other Adverse Events (participants affected / at risk) | 0/47 | 0/42 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Patients With Cardiac Arrhythmia Undergoing Cryoballoon (N=47) | Adult Patients With Cardiac Arrhythmia Undergoing Radiofrequency (N=42) | Adult Patients With Cardiac Arrhythmia Undergoing Pulsed Field Ablation (N=12)
Prolongation of an existing hospitalization (Surgical and medical procedures) | 0 | 1 | 0 — Related to the standard of care procedure. Due to a prolongation of hospitalization, this event was considered as Serious Adverse Event.

LIMITATIONS AND CAVEATS:
Only a limited amount of data (30 seconds) could be exported from the LS Pro system, which limited the correlation to only search a narrow region around the exported EGM data.

The data obtained from the PFA procedures could not be assessed due to incompatibility with the PVI Analyzer algorithm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT05043883/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT05043883/SAP_001.pdf
  • Informed Consent Form (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT05043883/ICF_002.pdf